CLINICAL TRIAL: NCT05262218
Title: A Phase IIa, Randomized, Double Blind, Placebo Controlled Study to Assess the Effect of PBF-680 in Patients With Moderate to Severe COPD on Top of the Standard Medication
Brief Title: Therapeutic Effect of PBF-680 in Patients With COPD
Acronym: Respire
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palobiofarma SL (Industry)
Collaborators: Scope International AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBF680CT-06
Record Dates: First submitted 2022-02-17; First posted 2022-03-02 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBF-680 (Experimental): PBF-680 is an Adenosine A1 receptor antagonist formulated in oral gelatine capsules
  Interventions: Drug: PBF-680 10mg
- Placebo (Placebo Comparator): Placebo formulated in oral gelatine capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PBF-680 10mg — PBF-680 10mg administered orally once a day
  Arms: PBF-680
Drug: Placebo — Placebo administered orally once a day
  Arms: Placebo

SUMMARY:
The purpose of the study is to investigate the effect of PBF-680 on the chronic inflammation and the lung function of patients with COPD on top of the standard medication. The effects of PBF-680 administration will also be examined with regards to symptom improvement and safety measures.One oral dose of PBF-680 or placebo will be administered daily for 4 weeks after randomization. The treatments will be administered double-blind with the Investigator and patient unaware of the treatment identity. A total of 102 COPD patients, either male or female, aged 40 to 80 years (inclusive) will be randomized.

DETAILED DESCRIPTION:
This is a Phase IIa, randomized, double-blind, placebo-controlled, parallel-group study to investigate the effect of the oral adenosine A1 receptor antagonist PBF-680 in patients with moderate to severe COPD over 4 weeks on top of the standard medication. It is planned to enroll approximately 114 patients at 8 sites with a target of 102 participants completing 4 weeks of treatment and key study assessments. The study comprises 5 visits: screening (Visit 1), randomization (Visit 2), 15 days-treatment visit (Visit 3), end of study visit (Visit 4) and follow up visit (visit 5).

Patients will be screened for eligibility (Visit 1). After the screening visit, patients will be instructed to continue at the same COPD standard medication (long-acting bronchodilators (long acting beta2-agonists [LABA] and/or long-acting muscarinic antagonists [LAMA]) and inhaled corticosteroids. Albuterol/salbutamol may be used as needed but must be held for at least 8 hours before a study visit.

Eligible patients will then return for Visit 2. The pre-dose FEV1 must be within 20% and 400ml of the predose FEV1 at the screening visit. Patients will be assessed for inclusion into the study, and if appropriate will be randomized to one of the two treatment arms. They will receive the first dose of study medication (PBF-680 or placebo) in the clinic (morning on fasting conditions) and have 3 spirometry performed in a timeframe of 3 hours. Patients will be discharged from the clinic, having been instructed to use the study medication on a once-a-day basis and in fasting conditions. The subject must record in a diary the daily self-administration of the study medication. The patient's diary will be provided together with the medication package dispensed on visit V2. The subject must be instructed to bring the medication package with all blisters to the site on visits V3 and V4.

Patients will return for 1 interim visit (Visit 3). At this visit, patients will bring the study medication pack containing the empty blisters and unused study medication. The dose of the study medication will be administered in the clinic. Spirometries will be performed at predose and 3h hour post dose.

At the final study visit (Visit 4), patients will be resident at the study center from the morning until at least 3 hours after dosing to allow for monitoring of lung function and study closeout procedures.

A follow-up visit (Visit 5) will occur 2 weeks after the final study visit as a safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Sign an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Male or female aged between 40 and 80 years inclusive, at the time of informed consent.
* Have a 12-lead ECG recording at screening (Visit 1) showing the following (and no changes at Visit 2 deemed clinically significant by the Investigator):

Heart rate between 50 and 90 beats per minute QT interval corrected for heart rate using Fridericia's formula (QTcF) interval ≤ 450 msec for males and ≤ 470 msec for females. QRS complex ≤ 120 msec PR interval ≤ 200 msec

* No clinically significant abnormality including morphology (e.g. left bundle branch block, atrioventricular nodal dysfunction, ST segment abnormality consistent with ischemia).
* Capable of complying with all study restrictions and procedures.
* Body mass index (BMI) between 20 and 35 kg/m2 (inclusive)
* COPD diagnosis: Patients with a clinical diagnosis of COPD as defined by Global Initiative for Chronic Obstructive Lung Disease - GOLD 20201 with symptoms compatible with COPD for at least 1 year prior to screening (Visit 1).
* Background triple therapy (ICS + LABA + LAMA) or double therapy (ICS + LABA or ICS + LAMA) for 3 months prior to randomization with a stable dose of medication for ≥1 month prior to Visit 1.
* Patient with blood eosinophils >100 cells/µL
* Ability to perform acceptable and reproducible spirometry. Post- bronchodilator (albuterol/salbutamol four puffs) spirometry at screening (Visit 1) must demonstrate a:

Post-bronchodilator FEV1/FVC ratio ≤ 0.70 Post-bronchodilator FEV1 ≥ 30 % and: ≤ 75 % of predicted normal.

* Clinically stable COPD in the 4 weeks prior to screening (Visit 1) and randomization (Visit 2).
* Meet the concomitant medication restrictions and be expected to do so for the rest of the study.
* Current and former smokers with a smoking history of ≥ 10 pack years.

Exclusion Criteria:

* Participants who have not been Vaccinated against SARS-CoV-2 and after performing a diagnostic nucleic acid test at screening visit, this would produce a positive result
* Participants with a significant COVID-19 illness ≥ OMS-4 within 6 months of enrolment
* A history of life-threatening COPD including Intensive Care Unit admission and requiring intubation.
* COPD exacerbation requiring oral steroids in the 3 months prior to randomization (Visit 2).
* A history of one or more hospitalizations for COPD in the 3 months prior to screening (Visit 1).
* Lower respiratory tract infection treated with antibiotics within 1 months of randomization (Visit 2).
* Increased pre-BD FEV1 at randomization visit (V2) compared to Screening (V1) of ≥ 400 mL or ≥ 20% of V1 FEV1.
* Evidence of cor pulmonale or clinically significant pulmonary hypertension.
* Other respiratory disorders: Patients with a current diagnosis of asthma, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung diseases, known alpha-1 antitrypsin deficiency or other active pulmonary diseases.
* Previous lung resection or lung reduction surgery.
* Oral therapies for COPD (e.g., theophylline, and roflumilast) in 1 month prior to screening (Visit 1) and throughout the study.
* Pulmonary rehabilitation, unless such treatment has been stable for 4 weeks prior to Visit 1) and remains stable during the trial.
* A history of, or reason to believe a subject has, drug or alcohol abuse within the past 3 years.
* Received an experimental drug within 30 days or five half-lives of Visit 2, whichever is longer.
* Women who are pregnant or breast-feeding.
* Patients with a history of chronic uncontrolled disease including, but not limited to, endocrine, active hyperthyroidism, neurological, hepatic, gastrointestinal, renal, hematological, urological, immunological, or ophthalmic diseases that the Investigator believes are clinically significant.
* Documented cardiovascular disease: arrhythmias, unstable angina, recent or suspected myocardial infarction within 6 months prior to screening, congestive heart failure, a history of unstable or uncontrolled hypertension, or has been diagnosed with hypertension in last 3 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the blood eosinophil count | 28 days
  Absolute and relative change from baseline (pre-dose ) will be computed. Mean difference will be provided.

SECONDARY OUTCOMES:
Effect of PBF-680 on trough forced expiratory volume in 1 second (FEV1) | 28 days
Change from baseline in prebronchodilator FEV1 at 3h post administration | 28 days
Change from baseline in postbronchodilator FEV1 at 3h post administration | 28 days
Change from baseline in the StGeorge's Respiratory Questionnaire (SGRQ-C) | 28 days
  St George's Respiratory Questionnaire Questionnaire is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. it is of 50 items questionnaire divided in two parts Part I (Symptoms): several scales; Part II (Activity and Impacts): dichotomous (true/false) Scores range from 0 to 100, with higher scores indicating more limitations.
Change from baseline in the Baseline Dyspnea Index (BDI)/ Transition Dyspnea Index (TDI) (BDI/TDI) | 28 days
  The Baseline Dyspnea Index is scored from 0 to 12 and is only assessed at baseline. The lower the score the worse the dyspnea severity. The Transition Dyspnea Index measures the change in dyspnea severity from the baseline as measured by the Baseline Dyspnea Index. It is rated by seven grades ranging from -3 (major deterioration) to +3 (major improvement).
Change from baseline in the COPD Assessment Test (CAT) | 28 Days
  The COPD Assessment Test (CAT) is questionnaire assessing globally the impact of COPD (cough, sputum, dysnea, chest tighteness) on health status. Number of items: 8 (one question assessing impact on sleep). Scaling of items:1 to 5. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life. No target score represents the best achievable outcome.
Change from baseline in the Modified Medical Research Council (MRC) breathlessness scales. | 28 days
  The Modified Medical Research Council(MRC) uses a simple grading system to assess a patient's level of breathlessness. It is rated by 4 grades ranging from 0 (best condition) to 4 (worse condition)
Number of subjects with treatment-related adverse events as assessed by CTCAE v4 | 28 days
  Adverse events will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4

CONTACTS AND LOCATIONS:
Overall Officials: Nahomi Castro Palomino, PhD, Study Chair — Palobiofarma S.L
Locations (7):
- Spain (7):
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Bellvitge, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital German Trias i Pujol, Barcelona
  - Hospital Sant Pau, Barcelona
  - Hospital Vall d´hebron, Barcelona

IPD SHARING:
Plan to Share IPD: No